CLINICAL TRIAL: NCT03218280
Title: Oxidative Stress Expression and Metabolic Imbalance in Critically Ill Polytrauma Patients and the Implications of Antioxidant Therapy on Clinical Outcomes
Acronym: OSPOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Romanian Society of Anesthesia and Intensive Care (Other)
Collaborators: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Responsible Party: Principal Investigator, Alexandru Florin Rogobete, Principal Investigator, Romanian Society of Anesthesia and Intensive Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20161212CA
Record Dates: First submitted 2017-04-03; First posted 2017-07-14 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Oxidative Stress; Polytrauma
Keywords: trauma; antioxidant; oxidative stress; Vitamin C; Ascorbic Acid
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antioxidant Therapy (Active Comparator)
  Interventions: Drug: Vitamin C
- Antioxidant Free (No Intervention)

INTERVENTIONS:
Drug: Vitamin C
  Arms: Antioxidant Therapy

SUMMARY:
Critically ill polytrauma patients have a number of physiological disorders secondary to trauma, such as systemic inflammatory response (SIRS), adult respiratory distress syndrome (ARDS), sepsis, oxidative stress (OS), and finally the multiple organ dysfunction syndrome (MODS). Another important aspect in terms of clinical outcome is the energy-metabolic status. Numerous studies have shown that implementing antioxidant therapy, capable of reducing the expression of pro-oxidative, pro-inflammatory and energetic-metabolic status, the mortality rate in critical patients decreases statistically significant. In this research paper, will be implemented a multimodal monitoring protocol that covers the use of biochemical, genetics and epigenetics biomarkers and the use of non-invasive medical devices to assess and monitor critical polytrauma patient. Also will be optimized the antioxidant treatment plan according to the needs of each patient.

DETAILED DESCRIPTION:
1. Objectives The project aims the integration for the first time in Romania of modern monitoring equipment for pro-oxidative, pro-inflammatory status and the energetic-metabolic necessary specific to the departments of anesthesia and intensive care, the clinical and laboratory data, genetic / epigenetic analyzes and existing information for the modulation and optimization of the intensive care for polytrauma patients. This way, the prospect of developing a decision support module for doctors to improve indices of mortality and morbidity in this area will be created. Reducing mortality and increasing quality of care is possible by providing a modern and complex monitoring system for critically ill polytrauma patient followed essentially by the acquisition, interpretation and synthesis in time of these biological signals and correlation with other clinical and laboratory data useful in modulating intensive care.

   The general objectives are to develop new areas of research in accordance with the trends of international research and with the economic and social romanian and european requirements by creating a integrated, innovative protocol with the improvement in the indices of mortality and morbidity in the intensive care of trauma patient through multimodality monitoring procedures and modulating intensive care management continuously in order to improve the public health system.

   The specific objectives of the study are the integration of modern methods for monitoring and optimizing therapeutic management depending on the individual patient (individualized management of intensive care); calculating severity and risk scores, both in the first 24 hours and continuously, providing medical decision support tools in real time; developing in an ergonomic, dynamic and standardized for viewing local and remote way the intensive care protocol modulated after modern techniques for non-invasive monitoring and cost-effective in the long term.

   Advantages of multimodal monitoring of pro-oxidative, pro-inflammatory and energetic-metabolic status through conventional laboratory analyzes, genetic / epigenetic analyzes and indirect calorimetry is represented by the particularly low time for obtaining the results, but also the pool of information brought on regarding the clinical status of these patients. Moreover, secondary it is possible to implement an intensive care that is modulated individually that reflects both on clinical outcome of the patient and the costs. Not least by obtaining a genetic array of specific pathophysiology's polymorphisms (SIRS, sepsis, ARDS, MODS) early and targeted therapies can be implemented that can significantly reduce mortality rates.
2. Impact The direct beneficiaries of the study are represented by physicians Department of Anesthesia and Intensive Care County Hospital Emergency "Pius Brinzeu" Timisoara that will have a very useful tool in clinical practice and research with direct impact on patient outcomes (approx. 3000 patients / year). Also, the entire local medical and scientific community: doctors, medical researchers and teachers. Through interdisciplinary nature of the specialty of anesthesia and intensive care, direct beneficiaries of research results in this area are represented by physicians from a wide range of medical specialties: surgery, neurosurgery, cardiology, infectious diseases, orthopedics and traumatology, clinical biology, genetics and so on. They will retrieve new information brought by research, will implement and apply it themselves on a new target groups of patients, thus expanding the distribution area of potential beneficiaries. Lastly, the economic environment through technology transfer from research results to other clinical and experimental centers.

   The indirect beneficiaries are represented by patients who will benefit directly from the implementation of the clinical trial results of research in anesthesia and intensive care: patients from clinics in the country and possibly abroad. Local and regional community - by improving the quality of medical services for the community, increased quality of life and level of economic and social reintegration of former patients. Local administration by savings from the local budget allocated to health with the implementation of new techniques and thus through reducing hospitalization time in the intensive care unit of these patients.
3. Statistical analysis Statistical analyzes will be carried out with specially designed computer equipment such as Prism 6 for Mac OSX v.6.0 (GraphPad Software, Inc., San Diego, CA) and Microsoft Office Excel (Microsoft Corporation, Bucharest, Romania). Statistical analysis of data recorded in the database will be to calculate frequencies and percentages for quantitative variables. Also, for the quantitative variables, the results will be expressed as the mean and standard deviation. Statistical comparisons used for test environments will be calculated with the unpaired t-test and for statistical comparisons used percentages using Chi square test. Statistical significance will be defined at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* ISS > 16
* age >18 y

Exclusion Criteria:

* refused to be enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Implications of Vitamin C on level of oxidative stress | Every 24 hours
  Change in baseline inflammatory biomarkers including Lipid expression modifications (HDL, LDL, Triglycerides, Cholesterol, mg%). Inflammation biomarkers (IL-6, Fibrinogen mg%) Protein expression (Total Proteins, Albumins, g) at every 24 hours following first administration of study drug, until the discharge form ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Rogobete, MSc, PhDs, Clinical Researcher, Principal Investigator — Emergency County Hospital Pius Brinzeu, Clinic of Anesthesia and Intensive Care; Ovidiu Bedreag, MD, PhD, Assist Prof, Study Director — Victor Babes University of Medicine and Pharmacy Timisoara; Dorel Sandesc, MD, PhD, Prof, Study Chair — Romanian Society of Anesthesia and Intensive Care

IPD SHARING:
Plan to Share IPD: Undecided